CLINICAL TRIAL: NCT03732300
Title: Evaluation of ASSIP - Attempted Suicide Short Intervention Program: a Randomized Controlled Trial
Brief Title: Attempted Suicide Short Intervention Program: a Randomized Controlled Trial
Acronym: EASI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Sebastian Olbrich, Deputy Head of Center for Social Psychiatry, University of Zurich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EASI
Record Dates: First submitted 2018-11-01; First posted 2018-11-06 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Suicidality; Suicide, Attempted
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted

STUDY DESIGN:
Intervention Model Description: Monocenter, open-label, randomized parallel two study arms (ASSIP vs control)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASSIP + TAU goup (Experimental): ASSIP psychotherapy intervention + treatment as usual (TAU)
  Interventions: Other: ASSIP
- TAU (No Intervention): Treatment as usual

INTERVENTIONS:
Other: ASSIP — Three PSychotherapy Sessions plus after 3/6/9/12 months individualized letters
  Other Names: Attempted Suicide Short Intervention Program
  Arms: ASSIP + TAU goup

SUMMARY:
"Attempted Suicide Short Intervention Program" (ASSIP) is a brief psychotherapy intervention after suicide attempts in psychiatric patients. The study aims to analyse the efficacy in a controlled trial by comparing number of patients with suicide attempts in a control group with treatment as usual and an intervention group with treatment as usual and ASSIP intervention.

Further, the study aims at indentifying electrophysiological, sociodempgraphical or smartphone-derived parameters for prediction of further suicide attempts.

DETAILED DESCRIPTION:
Suicide is the second leading cause of death among the 14-40 years old in Switzerland. Every year around 800'000 people all over the world die due to suicide (WHO, 2017). Preceding suicide attempts and self-harming behaviour have been found to be the main risk factor for completed suicide. The "Attempted Suicide Short Intervention Program" (ASSIP) has been designed to reduce further suicide attempts and suicide in patients after a suicide attempt. This study aims to replicate the findings of another study (Gysin-Maillart, Schwab, Soravia, Megert, & Michel, 2016) that show the efficacy of ASSIP. Further, it is intended to identify predictors for positive treatment outcome, i.e. a reduction of further suicide attempts in patients that had already committed a suicide attempt.

Main objective:

Assessment of efficacy of ASSIP by comparison of the number of patients that committed suicide attempts in the intervention (ASSIP) and the control group.

Secondary objectives:

• Identification of sociodemographic, clinical, electrophysiological and smartphone-based marker predicting the treatment outcome, rehospitalization rates and treatment costs Identification of predictors of treatment efficacy of ASSIP (by means of electroencephalogram parameters, electrocardiogram parameters, sensing app parameters, sociodemographic parameters and voice/video material parameters.

Identification of electrophysiological representations of suicidality (patient group, control group, healthy controls).

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Age 18 or older
* Attempted suicide no longer than 6 months before inclusion
* Treatment in and outpatient clinic of the University Hospital of Psychiatry Zurich, a daycare clinic or on a ward of the University Hospital of Psychiatry Zurich
* Able and willing to comply with all study requirements, especially being able to participate and understand psychotherapy sessions

Exclusion Criteria:

* Acute psychosis with delusion and/or hallucination
* Dementia
* Insufficient ability to communicate in German language
* Chronic self-harming behaviour without a direct intention of suicide (Wolfersdorf & Etzersdorfer, 2011)
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Current electroconvulsive therapy (do to interference between cognitive side effects and psychotherapeutic intervention)
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
suicide/attempted suicide | 12 months
  number of patients with attempted suicide or suicide

SECONDARY OUTCOMES:
Number of toal suicide attempts | 3,6,12 months
  Number of suicide attempts after 3/6 months/ one year (not a binary measure, each new attempt counts)
Hospitalization rates | 12 months
  Hospitalization rates and days and approximated treatment costs after one year
EEG-vigilance | baseline
  Electrophysiological wakefulness regulation as assessed via "VIGALL" algorithm in responders and non-responders
ECG Heart Rate Variability | baseline
  Electrophysiological heart rate variability (Total Power) associated with suicidality

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Olbrich, Principal Investigator — Department for Psychiatry, Psychotherapy and Psychosomatics, University Zurich
Locations (1):
- Department for Psychiatry, University Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gysin-Maillart A, Schwab S, Soravia L, Megert M, Michel K. A Novel Brief Therapy for Patients Who Attempt Suicide: A 24-months Follow-Up Randomized Controlled Study of the Attempted Suicide Short Intervention Program (ASSIP). PLoS Med. 2016 Mar 1;13(3):e1001968. doi: 10.1371/journal.pmed.1001968. eCollection 2016 Mar. PMID 26930055
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617